CLINICAL TRIAL: NCT01669928
Title: Hellenic Anglo Research Into Morning Or Evening Antihypertensive Drug deliverY Trial
Brief Title: Anti-hypertensive Medication Dosing Regimen in Effective Blood Pressure Control
Acronym: HARMONY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRO1749
Record Dates: First submitted 2012-07-02; First posted 2012-08-21 (Estimated); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evening medication (Active Comparator): Anti hypertensive medication in the evening (between 18.00 and 23.00)
  Interventions: Drug: Anti-hypertensive Medication -
- Morning medication (Active Comparator): Antihypertensive medication in the morning(between 06.00 and 11.00)
  Interventions: Drug: Anti-hypertensive Medication -

INTERVENTIONS:
Drug: Anti-hypertensive Medication - — Patients will be taking their routine blood pressure lowering medication prescribed by their GP, different patients will be using different blood pressure lowering medication.
  Dosing regimen either in the morning (between 06.00 and 11.00) or in the evening (between 18.00 and 23.00).
  Other Names: PR1 Diruetics; PR3 Beta Blockers; PR4 Calcium channel blockers; PR5 ACE inhibitors; PR6 Angiotensin II Receptor Blockers; PR7 Centrally acting agents; PR8 Alpha blockers; PR9 Direct Renin Inhibitors; PR10 Vasodilators

SUMMARY:
A randomised crossover trial of anti-hypertensive medication dosing regimen in effective blood pressure control.

To investigate whether there is a difference in 24 hour blood pressure (BP) control when antihypertensive medications are taken in the morning compared with the evening.

DETAILED DESCRIPTION:
The identification of any significant difference could lead to more effective therapeutic management of arterial hypertension, which in turn would result in a reduced cardiovascular burden, lower costs and a better quality of life for hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian patients aged 18-80 years;
* History of any grade of hypertension for at least 1 year, including at least 3 months of constant antihypertensive medication (consisting of ≥ 1 antihypertensive drugs, each administered in one dose daily), with reasonably controlled BP (≤150/90 mmHg and ≥ 115/75 mmHg on usual medication) based on previous clinic records, in the last 3 months.

Exclusion Criteria:

* BP levels > 150/90 mmHg or < 115/75 mmHg in the last 3 months.
* Postural hypotension, defined as symptoms resulting from a > 20 mm Hg drop of systolic BP or a > 10 mm Hg drop of diastolic BP or both between 1 and 3 min after standing from the sitting position.
* Known Extreme dippers at baseline (fall of mean night time SBP > 20% of mean day time SBP)
* Individuals with jobs which require night-time shift work.
* Pregnant women or those planning to become pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Poulter, MRCS LRCP MBBS MRCP MSc FRCP, Principal Investigator — Imperial College London
Locations (2):
- Aristotle University of Thessaloniki, Thessaloniki, Greece
- Imperial Clinical Trials Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemmer B. Clinical chronopharmacology: the importance of time in drug treatment. Ciba Found Symp. 1995;183:235-47; discussion 247-53. doi: 10.1002/9780470514597.ch13. PMID 7656688
- [Background] Bruguerolle B. Chronopharmacokinetics. Current status. Clin Pharmacokinet. 1998 Aug;35(2):83-94. doi: 10.2165/00003088-199835020-00001. PMID 9739478
- [Background] Rothwell PM, Howard SC, Dolan E, O'Brien E, Dobson JE, Dahlof B, Sever PS, Poulter NR. Prognostic significance of visit-to-visit variability, maximum systolic blood pressure, and episodic hypertension. Lancet. 2010 Mar 13;375(9718):895-905. doi: 10.1016/S0140-6736(10)60308-X. PMID 20226988
- [Background] Smolensky MH, Hermida RC, Ayala DE, Tiseo R, Portaluppi F. Administration-time-dependent effects of blood pressure-lowering medications: basis for the chronotherapy of hypertension. Blood Press Monit. 2010 Aug;15(4):173-80. doi: 10.1097/MBP.0b013e32833c7308. PMID 20571367
- [Background] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Influence of circadian time of hypertension treatment on cardiovascular risk: results of the MAPEC study. Chronobiol Int. 2010 Sep;27(8):1629-51. doi: 10.3109/07420528.2010.510230. PMID 20854139
- [Background] Heart Outcomes Prevention Evaluation Study Investigators; Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000 Jan 20;342(3):145-53. doi: 10.1056/NEJM200001203420301. PMID 10639539
- [Background] Mayet J, Chapman N, Li CK, Shahi M, Poulter NR, Sever PS, Foale RA, Thom SA. Ethnic differences in the hypertensive heart and 24-hour blood pressure profile. Hypertension. 1998 May;31(5):1190-4. doi: 10.1161/01.hyp.31.5.1190. PMID 9576134
- [Derived] Poulter NR, Savopoulos C, Anjum A, Apostolopoulou M, Chapman N, Cross M, Falaschetti E, Fotiadis S, James RM, Kanellos I, Szigeti M, Thom S, Sever P, Thompson D, Hatzitolios AI. Randomized Crossover Trial of the Impact of Morning or Evening Dosing of Antihypertensive Agents on 24-Hour Ambulatory Blood Pressure. Hypertension. 2018 Oct;72(4):870-873. doi: 10.1161/HYPERTENSIONAHA.118.11101. PMID 30354703

RESULTS

PARTICIPANT FLOW:
Groups:
- Morning Medication, Then Evening: Antihypertensive medication in the morning (between 06.00 and 11.00) for 6 months, then cross over to antihypertensive medication in the evening (between 18.00 and 23.00) for 6 months.
  Anti-hypertensive Medication -: Patients will be taking their routine blood pressure lowering medication prescribed by their GP, different patients will be using different blood pressure lowering medication.
- Evening Medication, Then Morning: Anti hypertensive medication in the evening (between 18.00 and 23.00) for 6 months, then cross over to antihypertensive medication in the morning (between 06.00 and 11.00) for 6 months,
  Anti-hypertensive Medication -: Patients will be taking their routine blood pressure lowering medication prescribed by their GP, different patients will be using different blood pressure lowering medication.
Period: First Intervention
Arm/Group | Morning Medication, Then Evening | Evening Medication, Then Morning
Started | 51 | 52
Completed | 48 | 47
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 5
Period: Second Intervention
Arm/Group | Morning Medication, Then Evening | Evening Medication, Then Morning
Started | 48 | 47
Completed | 48 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morning Medication, Then Evening | Evening Medication, Then Morning | Total
Number analyzed (Participants) | 51 | 52 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (11) | 62.8 (9.7) | 61.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 27 | 31 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 51 | 52 | 103
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 26 | 27 | 53
  Greece | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Changes in 24 Hour Systolic Blood Pressure
Description: Changes in 24 hour systolic Blood Pressure using ABPM
Time Frame: 6 months
Population: Total of 8 withdrawals / drop outs
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Morning Medication: Antihypertensive medication in the morning (between 06.00 and 11.00)
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 95
mm Hg | 129.65 (10.66) | 129.75 (12.75)

2. Secondary Outcome: Mean Day-time ABPM Systolic BP
Time Frame: 6 months
Population: Total of 8 withdrawals / drop outs
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 97
mm Hg | 132.24 (10.86) | 132.77 (12.87)

3. Secondary Outcome: Mean Day-time ABPM Diastolic BP
Time Frame: 6 months
Population: Total of 8 withdrawals / drop outs
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 97
mm Hg | 79.27 (7.73) | 80.55 (8.51)

4. Secondary Outcome: Μean Night Time ABPM Systolic BP
Time Frame: 6 months
Population: Total of 8 withdrawals / drop outs
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 97
mm Hg | 122.76 (12.18) | 121.08 (14.92)

5. Secondary Outcome: Μean Night Time ABPM Diastolic BP
Time Frame: 6 months
Population: Total of 8 withdrawals / drop outs
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 97
mm Hg | 70.92 (9.68) | 70.57 (9.67)

6. Secondary Outcome: Mean Clinic - Systolic BP
Description: This measure was assessed at a clinic.
Time Frame: 6 months
Population: Total of 8 withdrawals / drop outs
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 97
mm Hg | 129.37 (11.21) | 129.81 (12.53)

7. Secondary Outcome: Mean Clinic - Diastolic BP
Description: This measure was assessed at a clinic.
Time Frame: 6 months
Population: Total of 8 withdrawals / drop outs
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 97
mm Hg | 77.26 (7.12) | 77.41 (8.36)

8. Secondary Outcome: Self Reported Side Effects
Description: Serious Adverse Events reported during the trial
Time Frame: 12 months
Measure: Number; unit: Serious Adverse Events
Groups:
- Morning Medication: Antihypertensive medication in the morning (between 06.00 and 11.00) for 6 months
  Anti-hypertensive Medication -: Patients will be taking their routine blood pressure lowering medication prescribed by their GP, different patients will be using different blood pressure lowering medication.
- Evening Medication: Anti hypertensive medication in the evening
  Anti-hypertensive Medication -: Patients will be taking their routine blood pressure lowering medication prescribed by their GP, different patients will be using different blood pressure lowering medication.
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 97
Serious Adverse Events | 0 | 3

9. Secondary Outcome: Quality of Life Score
Description: Quality of Life Score via questionnaire - EQ-5D-5L Score scale is 0-100, 100 optimal health state.
Time Frame: 6 months
Population: Total of 8 withdrawals / drop outs
Measure: Mean (Standard Deviation); unit: Score out of 100
Arm/Group | Morning Medication | Evening Medication
Number analyzed (Participants) | 95 | 97
Score out of 100 | 84.14 (11.45) | 84.04 (10.25)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Morning Medication | Evening Medication
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/95 | 3/97
Other Adverse Events (participants affected / at risk) | 0/97 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morning Medication (N=95) | Evening Medication (N=97)
Chest pain (General disorders) | 0 (0) | 1 (1)
Planned admission for ERCP with stent. (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope episode (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No